CLINICAL TRIAL: NCT06226870
Title: Assessment of Vital Pulp Therapy Outcome Versus Root Canal Treatment in Management of Mature Permanent Molars with Irreversible Pulpitis and Apical Periodontitis(A Randomized Double-Blinded Clinical Trial)
Brief Title: Outcome of NSRCT Versus VPT in Management of Teeth with Symptomatic Irreversible Pulpitis Associated with Apical Periodontitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Abdelaal Mohamed, Assistant lecturer of Endodontics, Aswan University, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSRCT versus VPT
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-03

CONDITIONS: Endodontically Treated Teeth
MeSH Terms: conditions — Tooth, Nonvital | interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Computer will be used to generate a sequence of random numbers for the allocation of participants into the groups. Once the computer-generated randomization number will be obtained, it will be sealed in an opaque envelope by one of the investigators. After the clinical and radiographic findings, the envelope will be opened by a clinical assistant and treatment will be allocated to the patient based on the sequence generated. The patients will be blinded about the procedure, and a single operator will perform all the endodontic procedures after the informed written consent.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NSRCT Group (Experimental): Non-surgical root canal therapy
  Interventions: Procedure: root canal tretment
- VPT Group (Experimental): vital pulp therapy
  Interventions: Procedure: biodentin VPT
- VPT+PRF Group (Experimental): vital pulp therapy with PRF
  Interventions: Procedure: PRF

INTERVENTIONS:
Procedure: root canal tretment — traditional therapy
  Other Names: RCT
  Arms: NSRCT Group
Procedure: biodentin VPT — Alternative therapy
  Other Names: VPT
  Arms: VPT Group
Procedure: PRF — Alternative therapy
  Other Names: PRF plus VPT
  Arms: VPT+PRF Group

SUMMARY:
Pulpitis is the pulpal inflammation in response to irritants which are either microbial, chemical, or physical (mechanical and thermal) in origin. Clinically, pulpitis is termed as reversible or irreversible, whereas histologically, it is described as acute, chronic or hyperplastic . Pulpitis is considered reversible when the pulp can heal following conservative management . For such cases, a coronal pulpotomy is considered as a definitive treatment option having 78% to 90% of success rate . In irreversible pulpitis (IP), the pulp is not capable of healing, thus it is treated traditionally complete pulpectomy.

DETAILED DESCRIPTION:
I- Intervention

* Diagnosis to reach definitive diagnosis of SIP (positive response to pulp sensibility test) associated with SAP (PAI score ≤ 3), a detailed history and clinical examination should be collaborated with the radiographic evidence (CBCT) of apical periodontitis.
* Endodontic procedures
* Anesthetic protocol:

Tooth will be anaesthetized using 3.6 ml of 2% lidocaine with 1:100,000 epinephrine.

Inferior alveolar nerve block (IANB) supplemented by buccal infiltration will be accomplished using a standard aspirating syringe and a 27-G, long needle (C-K ject, CK Dental, Korea).

Access cavity preparation:

After rubber dam isolation, the tooth surface will be cleaned with gauze soaked in 5.25% sodium hypochlorite before the procedure.

All undermined tooth structure and caries will be removed with a diamond bur (komet, komet Dental, Germany) mounted on a high-speed handpiece.

Conventional access cavity will be performed by using round diamond bur (komet, komet Dental, Germany) for initial penetration. While Endo-Z (Prima Dental Group, UK) will be used for wall refinement to establish a straight-line access to canal orifices.

Preparation of the pulp chamber:

Immediately after access cavity preparation, any pulp tissue in the pulp chamber will be eliminated followed by cleansing with full concentration of sodium hypochlorite (6% NaOCl).

NSRCT group

* Patency Root canal patency will be established using a stainless-steel ISO size 10 K file (M. access, Dentsply, Switzerland).
* Working length determination The working length will be determined using an electronic apex locater (Tri Auto-ZX, J Morita, Japan) and re-confirmed by a digital intraoral periapical radiograph.
* Glide path Micro glidepath will be established using a stainless-steel ISO size 10 and 15 K manual files followed by macro glidepath using ProGlider® glide path rotary File.
* Root canal preparation The canals will be instrumented using Pro Taper Next® rotary files mounted on a torque controlled endodontic motor , in a continuous rotation motion, while torque and speed will be adjusted according to manufacturer instructions.
* Irrigation protocol During instrumentation Instrumentation will be supplemented with a copious irrigation of 2 ml of 6% NaOCl between each file and another delivered using a 30-gauge side-vented closed end irrigation neddle.

Final irrigation protocol An alternate use of 10 mL of 6% sodium hypochlorite and 10 mL of 17% EDTA for each canal, with an intermediate rinse with the same volumes of normal saline will be accomplished.

• Root canal obturation All canals will be dried using sterile paper points (ProTaper Next paper points .

Obturation will be done using a single cone technique with a bioceramic sealer .

VPT group All procedures will be carried out according to the guide-lines of the American Association of Endodontists (AAE) in 2021 for vital pulp therapy.

Haemostasis will be achieved with application of a cotton pellet moistened with 2.5% NaOCl for 2 min on which dry cotton pellet will be further placed. If required, the haemostasis will be carried out for another 6 minutes. In circumstances where the haemostasis still will not be achieved, the tooth will be excluded from the study.

Once the bleeding will be controlled, Biodentine will be mixed according to the manufacturer's instructions and will be placed in a 3-mm layer above the pulp tissue using an amalgam carrier and gently packed using a condenser . A layer of light-cure RMGIC will be placed over the pulpotomy agent and light-cured for 20s.

VPT with PRF group All procedures will be carried out according to the guide-lines of the American Association of Endodontists (AAE) in 2021 for vital pulp therapy.

Access cavity preparation and haemostasis will be carried out as mentioned previously, then PRF will be prepared by drawing the required amount of blood into a 10-mL test tube without an anticoagulant and centrifuged immediately using a table top centrifuge machine for 12 min. The resultant product consisted of the following three layers:

1. A cellular platelet poor plasma at the top of the tube.
2. Fibrin clot (PRF) in the middle of the tube.
3. Red blood corpuscles at the bottom of the tube. PRF will be obtained in the form of a membrane by squeezing out the fluids in the fibrin clot.

After that, the PRF membrane will be placed over the amputated pulp by using sterile tweezers. Biodentine will be will be placed in a 3-mm layer above the PRF gently packed using a condenser then a layer of light-cure RMGIC will be placed over the PRF and Biodentine then light-cured for 20s as mentioned in the previous group .

• Permanent restoration For all groups, the access cavity will be sealed with an appropriate post endodontic restoration within one week after root canal filling.

II. Outcome assessment:

Clinical evaluation and radiographic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (Category: American society of anesthesiologists class I) of either gender aged from 18-40 years.
* Permanent mature mandibular first molars with a definitive clinical diagnosis of SIP (positive response to pulp sensibility test) with SAP (PAI score ≤ 3)

Exclusion Criteria:

* Patients with systemic diseases such as (diabetes, hypertension, etc.…).
* Immunocompromised patients.
* Pregnant women and smokers.
* Patients with a history of antibiotic or analgesics intake within the few days before the intervention and cases with previously initiated endodontic treatment.
* Intraoperatively, where the haemostasis (application of 2.5% sodium hypochlorite pressure pack) could not be achieved within 10 minutes.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | at 24, 48 and 72-hours
  Preoperative and postoperative pain will be recorded on a point numeric rating scale by another operator. The numerical scale of pain is most commonly from 0 to 10, with 0 being "no pain" the lowest value and 10 being "the worst pain imaginable refer to the highest value, the lowest value means better outcome results.
Radiographic evaluation | at baseline ,6 and 12-months
  CBCT will be taken postoperatively to assess the periapical healing based on periapical index ( PAI) score. PAI score is ordinal scale of 5 scores ranging from 1 (healthy) lowest value to 5 (severe periodontitis with exacerbating features) highest value . The lowest value means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Abeer H Mahran, professor, Study Director — Ain Shams University
Locations (1):
- Faculty of dentistry, Minya, Egypt